CLINICAL TRIAL: NCT06835933
Title: Exploring Patterns in Postoperative Gastroesophageal Reflux Symptoms After Laparoscopic Sleeve Gastrectomy Based on the Presence of Preoperative Symptoms
Brief Title: Postoperative Gastroesophageal Reflux Symptoms After Laparoscopic Sleeve Gastrectomy Based on the Presence of Preoperative Symptoms
Status: Active, not recruiting | Type: Observational
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Sungsoo Park, Professor, Korea University Anam Hospital
Other Study IDs: SG-GERD
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-02

CONDITIONS: Obesity and Obesity-related Medical Conditions; Laparoscopic Sleeve Gastrectomy; Gastro-oesophageal Reflux
Keywords: obesity; diabetes mellitus; sleeve gastrectomy; gastro-esophageal reflux
MeSH Terms: conditions — Obesity; Gastroesophageal Reflux; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Preoperative symptom presence group: Patients whose preoperative symptom score from the modified GERD-HRQL questionnaire is not zero. For analyses of each symptom (heartburn and regurgitation), patients will be grouped based on the presence of the respective symptom: the heartburn symptom presence group for heartburn analysis and the regurgitation symptom presence group for regurgitation analysis.
  Interventions: Procedure: Laparoscopic sleeve gastrectomy
- Preoperative symptom absence group: Patients whose preoperative symptom score is zero, as assessed by the modified GERD-HRQL questionnaire. For each symptom analysis (heartburn and regurgitation), patients will be grouped based on the presence of the respective symptom: the heartburn symptom absence group for heartburn analysis and the regurgitation symptom absence group for regurgitation analysis.
  Interventions: Procedure: Laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Laparoscopic sleeve gastrectomy (LSG) is most commonly performed bariatric/metabolic surgery. LSG is performed in patients with obesity and/or obesity-related comorbidities. During LSG, the stomach was resected from 5 cm proximal to the pylorus to the angle of His, guided by a 36-French bougie. In patients with hiatal hernia, concomitant HHR was also performed with LSG using non-absorbable sutures. Routine oral potassium-competitive acid blocker (PCAB) was prescribed for 3 months after surgery and the discontinuation of PCAB was determined based on GERD symptoms at the 3-month visit.

SUMMARY:
This study aims to investigate the patterns of reflux symptoms after laparoscopic sleeve gastrectomy based on the presence or absence of preoperative gastroesophageal reflux symptoms.

DETAILED DESCRIPTION:
Obesity is a well-known risk factor for gastroesophageal reflux disease (GERD), and laparoscopic sleeve gastrectomy (LSG) is the most commonly performed bariatric/metabolic surgery. However, patients often experience reflux symptoms after LSG, and those with severe reflux symptoms or severe erosive esophagitis have been excluded from candidates for LSG. This study aims to analyze the patterns of postoperative reflux symptoms based on the presence of preoperative reflux symptoms.

Prospectively established databases of patients assessed for reflux symptoms at a single institution will be retrospectively reviewed. A total of 64 patients who underwent LSG between April 2020 and March 2023 will be included in this study. The modified GERD-HRQL (GERD- health-related quality of life) questionnaire was used to evaluate gastroesophageal reflux symptoms before LSG and at 1, 3, 6, 9, and 12 months after surgery. Reflux symptoms will be categorized into heartburn and regurgitation, and the patterns of heartburn and regurgitation scores included in the modified GERD-HRQL questionnaire will be analyzed. The patients will be classified based on the presence or absence of preoperative reflux symptoms, and the patterns of symptom scores within each group will be analyzed. We will also measure the correlation between whether hiatal hernia repair was performed with laparoscopic sleeve gastrectomy and adiposity-related parameters, including preoperative and postoperative body mass index (BMI), preoperative and postoperative waist circumference (WC), the percentage of total weight loss (%TWL), and the percentage of WC reduction, and changes in postoperative symptom scores.

ELIGIBILITY:
Inclusion Criteria:

1. patients with age greater than 19 years
2. patients who underwent laparoscopic sleeve gastrectomy from March 2019 to March 2023
3. patients with postoperative follow-up longer than one month after LSG
4. patients who answered preoperative and postoperative GERD questionnaire (Korean translated version of modified GERD-HRQL)

Exclusion Criteria:

1) patients with missing or incomplete postoperative GERD questionnaires

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent laparoscopic sleeve gastrectomy
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Symptom scores from the modified GERD-HRQL | before laparoscopic sleeve gastrectomy and at 1, 3, 6, 9, 12 months after surgery
  The modified GERD-HRQL consists of 15 questions with a 6-point Likert scale ranging from 0 to 5. Among these, six questions are related to heartburn, while another six focus on regurgitation. Symptom scores including heartburn and regurgitation scores were defined as the sum of the six questions related to each symptom.

SECONDARY OUTCOMES:
Hiatal hernia repair with laparoscopic sleeve gastrectomy (performed or not) | during laparoscopic sleeve gastrectomy
  In patients with hiatal hernia, hiatal hernia repair was performed with laparoscopic sleeve gastrectomy. A subgroup analysis will be conducted based on the presence or absence of a hiatal hernia.
  We will also analyze the correlation between whether hiatal hernia repair was performed with laparoscopic sleeve gastrectomy and the changes in postoperative symptom scores.
  * The changes in postoperative symptom scores = postoperative symptom scores - preoperative symptom scores
Adiposity-related parameters | before laparoscopic sleeve gastrectomy and at 1, 3, 6, 9, 12 months after surgery (WC: before laparoscopic sleeve gastrectomy and at 3, 6, 9, 12 months after surgery)
  We will analyze the correlation between adiposity-related parameters, including preoperative and postoperative body mass index (BMI), preoperative and postoperative waist circumference (WC), the percentage of total weight loss (%TWL), and the percentage of WC reduction, and the changes in postoperative symptom scores.
  * The changes in postoperative symptom scores = postoperative symptom scores - preoperative symptom scores; BMI = body weight (kg) / height (m)^2;
  * TWL = (preoperative body weight - postoperative body weight)/preoperative body weight x 100 (%); WC reduction = (preoperative WC - postoperative WC)/preoperative WC x 100 (%); ** WC was measured at the level of the umbilicus.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
According to private information law, the IPD generated and/or analyzed for this study will not be shared.

REFERENCES:
- [Background] Balla A, Leone G, Ribichini E, Sacchi MC, Genco A, Pronio A, Paganini AM, Badiali D. Gastroesophageal Reflux Disease - Health-Related Quality of Life Questionnaire: prospective development and validation in Italian. Eur J Gastroenterol Hepatol. 2021 Mar 1;33(3):339-345. doi: 10.1097/MEG.0000000000001914. PMID 32925505
- [Background] Velanovich V, Vallance SR, Gusz JR, Tapia FV, Harkabus MA. Quality of life scale for gastroesophageal reflux disease. J Am Coll Surg. 1996 Sep;183(3):217-24. PMID 8784314
- [Background] Eisenberg D, Shikora SA, Aarts E, Aminian A, Angrisani L, Cohen RV, de Luca M, Faria SL, Goodpaster KPS, Haddad A, Himpens JM, Kow L, Kurian M, Loi K, Mahawar K, Nimeri A, O'Kane M, Papasavas PK, Ponce J, Pratt JSA, Rogers AM, Steele KE, Suter M, Kothari SN. 2022 American Society of Metabolic and Bariatric Surgery (ASMBS) and International Federation for the Surgery of Obesity and Metabolic Disorders (IFSO) Indications for Metabolic and Bariatric Surgery. Obes Surg. 2023 Jan;33(1):3-14. doi: 10.1007/s11695-022-06332-1. PMID 36336720
- [Background] Kim MS, Lee I, Natarajan P, Do R, Kwon Y, Shin JI, Solmi M, Kim JY, Won HH, Park S. Integration of observational and causal evidence for the association between adiposity and 17 gastrointestinal outcomes: An umbrella review and meta-analysis. Obes Rev. 2024 Dec;25(12):e13823. doi: 10.1111/obr.13823. Epub 2024 Sep 4. PMID 39233338
- [Background] Silveira FC, Poa-Li C, Pergamo M, Gujral A, Kolli S, Fielding GA, Ren-Fielding CJ, Schwack BF. The Effect of Laparoscopic Sleeve Gastrectomy on Gastroesophageal Reflux Disease. Obes Surg. 2021 Mar;31(3):1139-1146. doi: 10.1007/s11695-020-05111-0. Epub 2020 Nov 26. PMID 33244654